CLINICAL TRIAL: NCT01200017
Title: An Expanded Access Study of the Feasibility of Using the CliniMACS® Device for CD34+ Cell Selection and T Cell Depletion for Graft-versus-Host Disease Prophylaxis in Alternative Donor Stem Cell Transplant Recipients
Brief Title: Expanded Access Protocol (EAP) Using the CliniMACS® Device for Pediatric Haplocompatible Donor Stem Cell Transplant
Status: No longer available | Type: Expanded Access
Sponsor: Christopher Dvorak (Other)
Responsible Party: Sponsor-Investigator, Christopher Dvorak, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Other Study IDs: 10082; NCI-2020-02478 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Myeloid Leukemia; Myelodysplastic Syndrome; Lymphomas; Bone Marrow Failure; Hemoglobinopathy; Immune Deficiency; Osteopetrosis; Cytopenias; Leukocyte Disorders; Anemia Due to Intrinsic Red Cell Abnormality
Keywords: T cell depleted; Matched unrelated donors; Haplocompatible donors; Graft vs Host Disease; Hemoglobinopathies; Leukemia; Leukemia, Lymphoid; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma; Myelodysplastic Syndromes; Preleukemia; Osteopetrosis; Pancytopenia; Immune System Diseases; Hematologic Diseases; Genetic Diseases, Inborn; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Myeloproliferative Disorders; Bone Marrow Diseases; Precancerous Conditions; Osteosclerosis; Osteochondrodysplasias; Bone Diseases, Developmental; Bone Diseases; Musculoskeletal Diseases; Severe acquired and congenital cytopenias; White and red blood cell abnormalities
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Lymphoma; Bone Marrow Failure Disorders; Hemoglobinopathies; Immunologic Deficiency Syndromes; Osteopetrosis; Cytopenia; Leukocyte Disorders; Graft vs Host Disease; Leukemia; Leukemia, Lymphoid; Leukemia, Myeloid; Preleukemia; Pancytopenia; Immune System Diseases; Hematologic Diseases; Genetic Diseases, Inborn; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Myeloproliferative Disorders; Bone Marrow Diseases; Precancerous Conditions; Osteosclerosis; Osteochondrodysplasias; Bone Diseases, Developmental; Bone Diseases; Musculoskeletal Diseases | interventions — Bone Marrow Transplantation

INTERVENTIONS:
Biological: CD34+ enriched, T Cell Depleted donor stem cell product — stem cell transplant
  Other Names: bone marrow transplant

SUMMARY:
This protocol provides expanded access to bone marrow transplants for children who lack a histocompatible (tissue matched) stem cell or bone marrow donor when an alternative donor (unrelated donor or half-matched related donor) is available to donate. In this procedure, some of the blood forming cells (the stem cells) are collected from the blood of a partially human leukocyte antigen (HLA) matched (haploidentical) donor and are transplanted into the patient (the recipient) after administration of a "conditioning regimen". A conditioning regimen consists of chemotherapy and sometimes radiation to the entire body (total body irradiation, or TBI), which is meant to destroy the cancer cells and suppress the recipient's immune system to allow the transplanted cells to take (grow). A major problem after a transplant from an alternative donor is increased risk of Graft-versus-Host Disease (GVHD), which occurs when donor T cells (white blood cells that are involved with the body's immune response) attack other tissues or organs like the skin, liver and intestines of the transplant recipient. In this study, stem cells that are obtained from a partially-matched donor will be highly purified using the investigational CliniMACS® stem cell selection device in an effort to achieve specific T cell target values. The primary aim of the study is to help improve overall survival with haploidentical stem cell transplant in a high risk patient population by limiting the complication of GVHD.

DETAILED DESCRIPTION:
Patients will be enrolled with alternative (mismatched/haplocompatible) related donors or unrelated donors either for an initial transplant or as a rescue following rejection of a previous graft or relapse following a previous transplant. For patients with mismatched related donors, the majority of clinical experience has been with a T cell-depleted PBSC product. Currently, no FDA-approved method for T cell depletion exists. Recent experience with the CliniMACS® device has produced excellent results with a 70-75% survival in children, many of whom were high risk patients.

Patients that receive transplants from unrelated donors usually receive stem cells that are not T cell-depleted. However, this is associated with a high risk of GVHD. The excellent results with mismatched related donor transplants justify expanding this approach to unrelated donor transplant recipients if the HLA mismatch is sufficiently great. It is anticipated that the use of the CliniMACS® device will result in a very low risk of GVHD without the need for post-transplant immunosuppression. The outcomes in relatively small studies for children receiving unrelated donor transplants using the CliniMACS® have been comparable to or better than those receiving T replete transplants with post-transplant immunosuppression.

This protocol will allow the use of patient-specific conditioning regimens. Some patients have contraindications to certain components of the conditioning regimen used for our ongoing study under BB-IND 8817 (CC# 01151). An example is a patient with pre-existing organ dysfunction that would be better served by the use of a reduced intensity conditioning regimen. Another example is a patient for whom total body irradiation is contraindicated due to very young age or prior radiation therapy. Finally, patients who would be otherwise eligible for the predecessor study but who do not have an eligible related donor or a closely matched unrelated donor would be eligible for this study. The target CD3+ T cell dose that will be given will be 3 x 10^4/kg. The University of California, San Francisco Protocol CC#01151 uses a dose of 3 x 10^4/kg. The T cell dose in the graft is usually < 1 x 10^4/kg after processing and T cells are added to the product.

ELIGIBILITY:
Inclusion Criteria:

* >2 months - 30 years
* Patient must have a malignant or non-malignant disease that can benefit from alternative stem cell transplantation according to standard practice guidelines for including patients for transplant as outlined in UCSF Pediatric Bone Marrow Transplant (BMT) Standard Operating Procedure (SOP) #206.04. Examples include acute and chronic leukemias, myelodysplastic syndrome, lymphoma, severe acquired and congenital cytopenias, white and red blood cell abnormalities, inborn errors of metabolism and immunodeficiencies. Patient with Fanconi's Anemia will be eligible regardless of match with donor.
* Patients with acute leukemia (AML excepted) or lymphoma must be in remission at the time of transplant.
* Patients must lack a healthy human leukocyte antigen (HLA)-identical related donor.
* Recipient or authorized guardian must sign informed consent for this study.
* If recipient is female and of child-bearing age, negative pregnancy test.
* Patient must have a healthy, willing mismatched related or an unrelated donor who is:

  * Able to receive Granulocyte colony-stimulating factor (G-CSF) +/- Plerixafor and undergo apheresis either through placement of catheters in antecubital veins or a temporary central venous catheter,
  * For Related donor: sibling, half-sibling, parent, cousin, aunt, uncle or grandparent will all be considered eligible.
  * For Related donor: HLA antigen genotypic match ≥ 4/8 and ≤ 7/8 (haplocompatible).
  * For unrelated donor: 6/8 or 7/8 HLA antigen match (if two mismatches, they must be at different loci).
  * Complete medical history, physical and screening for infectious diseases that are acceptable for donation.
  * If donor is female and of child-bearing age, negative pregnancy test.
  * Absence of anti-HLA antibodies in recipient directed against donor antigens.
  * Donor must be willing to sign informed consent for this study. If donor is < 18 years of age, donor must be willing to give assent and parents willing to sign informed consent.
* Be suitable for an autologous gene-modified transplant:

  * Using either bone marrow or cytokine-mobilized peripheral blood stem cells (PBSC).
  * Patient or authorized guardian must sign informed consent for this study.
* For unrelated donors: Per New Algorithm, Jan. 14, 2016, effective immediately, National Marrow Donor Program (NMDP) "Be The Match" is adopting a revised algorithm for determining if a donor is a research subject on their recipient's research protocol: The NMDP will inform the donor of the activities and the use of donor's apheresis product to be used in this study and obtain written consent from the donor. Transplant centers are sent documentation of the donor consent to participate in the research support activities. (The revised algorithm can be found on the "Be the Match Clinical Network")
* Criteria to consider when choosing among related haplo donors:

  * CMV positive donor is preferred over other factors. CMV negative donor can be used only if recipient is CMV negative.
  * HLA disparity i.e. 2 Ag mismatch preferred over 3 Ag mismatch; Drβ1 match preferred over class I match; HLA-C matched preferred over A and B match.
  * killer immunoglobulin-like receptor (KIR) mismatch in GVH direction is preferred for patients with malignant disorders
  * ABO compatibility
* Age ≥ 2 months

Exclusion Criteria:

* Patient with an anticipated life expectancy of < 1 month
* Active infectious hepatitis or cytomegalovirus (CMV) disease (organ involvement)
* Human immunodeficiency virus (HIV) or Human T-lymphotropic virus (HTLV-I/II) infection
* Cardiac ejection fraction < 45%; can be lower if patient is not in clinical cardiac failure and a reduced intensity conditioning regimen is used.
* Creatinine clearance <60 ml/min/1.72 m2; can be lower if a reduced intensity conditioning regimen is used.
* Pulmonary diffusion capacity (corrected for hemoglobin), forced expiratory volume in one second (FEV1), or forced vital capacity (FVC) <60% of predicted or oxygen saturation (O2 sat) > 94% on room air if unable to perform pulmonary function tests (PFTs); can be lower if a reduced intensity conditioning regimen is used.
* Serum alanine aminotransferase (ALT) > 5 x upper limit of normal (can be up to 10x upper limit of normal if a reduced intensity conditioning regimen is used) or bilirubin > 2.
* Performance score (Lansky/Karnofsky) < 50
* Any condition that compromises compliance with the procedures of this protocol, as judged by the principal investigator.

Ages: 2 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dvorak, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

DOCUMENTS (1):
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT01200017/Prot_000.pdf